CLINICAL TRIAL: NCT04534985
Title: Time Restricted Feeding in Overweight and Obese Adults With Autosomal Dominant Polycystic Kidney Disease
Brief Title: Time Restricted Feeding in Autosomal Dominant Polycystic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: PKD Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 20-1262
Record Dates: First submitted 2020-08-25; First posted 2020-09-01 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Polycystic Kidney, Autosomal Dominant
Keywords: Timed Feeding; Kidney Diseases; Body Weight
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant; Kidney Diseases; Body Weight | interventions — Diet

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Time Restricted Feeding (Experimental): Instructed to eat within an 8-hr window, beginning within 3 hrs of waking. In addition, provide current clinical recommendations for the management of ADPKD, as well as chronic kidney disease, including moderate dietary sodium restriction (2.3-3 g), appropriate hydration, protein intake of 0.8/1.0 g/kg ideal body weight, moderate daily phosphate restriction (800 mg), and moderation in caloric intake.
  Interventions: Behavioral: Dietary
- Healthy Eating Advice without Time Restricted Feeding (Active Comparator): Curriculum for the healthy eating control group will emphasize current clinical recommendations for the management of ADPKD, as well as chronic kidney disease, including moderate dietary sodium restriction (2.3-3 g), appropriate hydration, protein intake of 0.8/1.0 g/kg ideal body weight, moderate daily phosphate restriction (800 mg), and moderation in caloric intake.
  Interventions: Behavioral: Dietary

INTERVENTIONS:
Behavioral: Dietary — Dietary intake behavioral intervention via time restricted feeding and normal healthy eating recommendations vs. normal healthy eating recommendations without restricted

SUMMARY:
The proposed research will determine the feasibility of a time restricted feeding intervention,a fasting regimen that restricts eating to a feeding window (8 hrs/day) for 1 year in adults with autosomal dominant polycystic kidney disease (ADPKD) who are overweight or obese. The study will provide valuable information on the intervention in terms of safety, adherence, acceptability, and tolerability. Last, this pilot trial will provide initial insight into biological changes including abdominal adiposity, changes in kidney growth and function, and markers of biological pathways related to the intervention.

DETAILED DESCRIPTION:
Mounting evidence suggests that a metabolic defect exists in autosomal dominant polycystic kidney disease (ADPKD), which likely contributes to cystic epithelial proliferation and subsequent cyst growth. There are notable overlapping features and pathways among metabolism, obesity, and/or ADPKD. The investigators recently reported that in the Halt Progression of Polycystic Kidney Disease (HALT-PKD) Study A that overweight and obesity are strong independent predictors of more rapid kidney growth. Moving beyond body mass index, the investigators have novel preliminary data using magnetic resonance images (MRIs) from a small number of participants from HALT-PKD Study A that abdominal adiposity is an independent predictor of kidney growth and kidney function decline. Adipocytes do not simply act as a fat reservoir but are active endocrine organs that promote release of pro-inflammatory cytokines and produce adipokines. Numerous signaling pathways promoted by adipocytes are also implicated in cystogenesis. Periods of fasting may counter adiposity-mediated signaling pathways and slow ADPKD progression. Mild-to-moderate food restriction profoundly slows cyst growth and maintains renal function in rodent models of ADPKD, which are characterized by metabolic reprogramming favoring enhanced aerobic glycolysis. Notably, fasting promotes a shift from carbohydrate to fat metabolism, which could suppress cyst growth. The investigators are currently conducting an ongoing behavioral weight loss pilot trial (based on either daily caloric restriction or intermittent fasting) in adults with ADPKD who are overweight/obese. As an alternative to these approaches, time-restricted feeding (TRF) is a novel fasting regimen that restricts eating to a feeding window (typically 8-12 hrs/day). As isocaloric TRF reduces disease progression in a rodent model of ADPKD, including kidney: body weight and mammalian target of rapamycin (mTOR) activity, it may be an alternative and easier to adhere to dietary strategy to slow ADPKD progression. Specific Aim: Determine the feasibility of TRF without energy intake restriction in adults with ADPKD and overweight/obesity. The study will determine adherence to TRF by assessing the percent of participants achieving the goal of eating within an 8-hour TRF window, measured objectively with a photographic food record and verified with continuous glucose monitoring data. The study will also further assess the safety, acceptability, and tolerability of TRF by evaluation of safety labs, adverse events, and quality of life measures, as well as changes in abdominal adiposity and total kidney volume (TKV) by magnetic resonance imaging (MRI), and markers of biological pathways (AMP-activated protein kinase [AMPK], mTOR, insulin-like growth factor 1 [IGF1]).

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-65 years
2. ADPKD diagnosis based on the modified Pei-Ravine criteria
3. BMI 25-45 kg/m^2
4. Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) estimated glomerular filtration rate ≥30 mL/min/1.73 m^2
5. Access to the internet with video chat capabilities and smartphone
6. Typical eating duration >12 hrs/day
7. Not currently participating in another interventional study or weight loss program
8. Ability to provide informed consent

Exclusion Criteria:

1. Diabetes mellitus (diagnosis or fasting glucose >126 mg/dL or Hemoglobin A1C >6.5%)
2. Current nicotine use or history of use in the past 12 months
3. Alcohol or substance abuse (self-report or undergoing treatment)
4. History of hospitalization or major surgery within the last 3 months
5. Untreated dyslipidemia (low density lipoprotein cholesterol > 190 mg/dL or triglycerides >400 mg/dL)
6. Uncontrolled hypertension (systolic blood pressure > 160 or diastolic blood pressure >100 mm Hg)
7. Pregnancy, lactation, or unwillingness to use adequate birth control
8. Cardiovascular disease, peripheral vascular disease, cerebrovascular disease, significant pulmonary or gastrointestinal disease (described below), cancer (within the last 5 years, except skin cancer or other cancers considered cured with excellent prognosis)
9. Significant gastrointestinal disorders including: chronic malabsorptive conditions, peptic ulcer disease, Crohn's disease, ulcerative colitis, chronic diarrhea, or active gallbladder disease
10. Regular use of prescription or over-the-counter medications that may affect weight, appetite, food intake, or energy metabolism (e.g. appetite suppressants, lithium, stimulants, anti-psychotics, tricyclic antidepressants; study physician will be consulted as needed; antibiotics started during the intervention period are not an exclusion); regular use of obesity pharmacotherapeutic agents within the last 6 month
11. History of clinically diagnosed eating disorder including anorexia nervosa, bulimia, binge eating disorder. Score >20 on the Eating Attitudes Test (EATS)-2653 will require further assessment by the Study MD to determine if it is appropriate for the subject to participate in the study.
12. Weight loss >5% in past 3 months for any reason except post-partum weight loss; weight gain >5% in past 3 months requires assessment by PI to determine reason for weight gain and if it is appropriate for the subject to participate in the study.
13. Untreated hyper- or hyperthyroidism (TSH outside of normal range for laboratory or history of uncontrolled thyroid disorder). History of thyroid disorder or current thyroid disease treated with stable medication regimen for at least 6 months in acceptable.
14. Current severe depression or history of severe depression within the previous year, based on DSM-IV-TR criteria for Major Depressive Episode. Score > 18 on the Beck Depression Inventory will require further assessment by the Study MD to determine if it is appropriate for the subject to participate in the study.
15. History of other significant psychiatric illness (e.g. psychosis, schizophrenia, mania, bipolar disorder) which in the opinion of the Study MD would interfere with ability to adhere to dietary interventions.
16. Inability to cooperate with/clinical contraindication for MRI including severe claustrophobia, implants, devices, or non-removable body piercings

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2021-02-09 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Adherence | 1 year
  Percent adherence to the 8-hr TRF window (during the 7 day recordng period)
Feasibility to enroll participants | Through study enrollment, an expected duration of 12 months
  Numbers of individuals pre-screened and enrolled
Feasibility to retain participants | Through study completion, an expected duration of 24 months
  Numbers of individuals retained

SECONDARY OUTCOMES:
Safety and tolerability, measured as adverse events | Through study completion, an expected duration of 24 months
  Number of participants with treatment-related adverse events in each group as evaluated by the Safety Officer
Change in Body Weight | 1 year
  Body weight will be measured at baseline and monthly, using BodyTrace scales for remote, secure transmission of data.
Change in Abdominal adiposity | 1 year
  Abdominal adiposity will be quantified using MRI
Change in Body Composition | 1 year
  Body composition measured via dual-energy X-ray absorptiometry (DEXA)
Change in insulin-like growth factor binding protein-1 levels | 1 year
  Fasting serum insulin-like growth factor binding protein-1 (IGFBP-1) levels will be evaluated in each group
Change in serum insulin-like growth factor-1 levels | 1 year
  Fasting serum insulin-like growth factor-1 (IGF-1) levels will be evaluated in each group
Change in peripheral blood mononuclear cell (PBMC) AMPK expression | 1 year
  Peripheral blood mononuclear cell protein expression of AMP-activated kinase (AMPK) in each group
Change in PBMC S6K expression | 1 year
  Peripheral blood mononuclear cell protein expression of S6 kinase (S6K) in each group
Change in β-hydroxybutyrate levels | 1 year
  Serum β-hydroxybutyrate levels in each group
Change in total kidney volume by magnetic resonance imaging (MRI) | 1 year
  Change in total kidney volume by MRI in each group
Change in quality of life | 1 year
  Quality of life (QOL) will be assessed with the RAND 36 Item Health Survey (RAND-36) physical and mental health component summary score
Change in mood | 1 year
  Mood state will be assessed with the Profile of Mood States 2 (POMS-2)
Change in pain | 1 year
  Modified version of the Wisconsin Brief Pain Survey

OTHER OUTCOMES:
Change in resting energy expenditure | 1 year
  Standard indirect calorimetry
Change in energy intake | 1 year
  24-hr dietary recalls will be analyzed using a random day in the 7-day photographic food record/continuous glucose monitoring collection period to evaluate self-reported energy intake
Change in macronutrient intake | 1 year
  24-hr dietary recalls will be analyzed using a random day in the 7-day photographic food record/CGM collection period to evaluate self-reported energy intake
Change in self-reported physical activity | 1 year
  Self-reported physical activity will be quantified using the Stanford Physical Activity Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Nowak, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado - Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in ADPKD. Data shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements (i.e. data use agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, ICF
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA).

REFERENCES:
- [Derived] St Pierre K, Cashmore BA, Bolignano D, Zoccali C, Ruospo M, Craig JC, Strippoli GF, Mallett AJ, Green SC, Tunnicliffe DJ. Interventions for preventing the progression of autosomal dominant polycystic kidney disease. Cochrane Database Syst Rev. 2024 Oct 2;10(10):CD010294. doi: 10.1002/14651858.CD010294.pub3. PMID 39356039
- [Derived] Chebib FT, Nowak KL, Chonchol MB, Bing K, Ghanem A, Rahbari-Oskoui FF, Dahl NK, Mrug M. Polycystic Kidney Disease Diet: What is Known and What is Safe. Clin J Am Soc Nephrol. 2024 May 1;19(5):664-682. doi: 10.2215/CJN.0000000000000326. Epub 2023 Sep 20. PMID 37729939